CLINICAL TRIAL: NCT04328532
Title: MRI Screening of Placenta Adhesion Abnormalities
Acronym: DIANE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, BERTHOLDT Charline, Doctor, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-A02794-53
Record Dates: First submitted 2020-02-27; First posted 2020-03-31 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Placenta; Implantation

STUDY DESIGN:
Intervention Model Description: Prospective interventional clinical cohort study, monocentric, controlled, open.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pregnancy with risk factors for PPA (Experimental)
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — MRI examination (45 min max) with potential oxygen delivery for 10 min

SUMMARY:
Placenta Adhesion Abnormalities (PAA) are the consequence of an excessive invasion of the placenta within the myometrium. PAA are related to severe maternal pregnancy outcomes, especially in case of incidental discovery during delivery that increase the risk of intraoperative massive bleeding, hysterectomy and even maternal death. Ultrasound is the standard modality for diagnosing PAA, but Magnetic Resonance Imaging (MRI) has been increasingly performed in the case of inconclusive sonographic findings. However, standard morphological MRI sequences appear as insufficient to improve the sensitivity and specificity values for detecting PAA, while quantitative MRI may be more efficient.

The main objective of this study is to characterize the diagnostic performance of quantitative MRI parameters (mainly Apparent Diffusion Coefficient, T2 and T2*) reflecting placental perfusion and/or oxygenation at high field, without injection of gadolinium-based agent, for the detection of PAA in women with ongoing pregnancy between 30 and 38 weeks of gestation with risk factors for PPA.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant participant between 30 and 38 weeks of gestation,
* Age ≥18 years old,
* Participant who completed the preliminary medical examination,
* Participant who has received full information about the organization of the research and has signed her informed consent.
* Participant planning to give birth at CHRU of Nancy
* Participant presenting risk factors for PAA : low-lying or covering placenta or in front of the uterine scar.

Exclusion Criteria:

* Multiple pregnancy,
* Participant presenting at least one contraindication or restriction to performing an MRI as described in the protocol, in accordance with the current recommendations,
* Participant unable to understand or follow study procedure,
* Person referred to in Articles L. 1121-6 to L. 1121-8, L1122-2 and L. 1122-1-2 of the Public Health Code.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2026-10-21 (Estimated); Study Completion 2026-10-21 (Estimated)

PRIMARY OUTCOMES:
Area under the ROC curve of the T2 relaxation time mean value | Through study completion, an average of 6 months
Area under the ROC curve of the T2* relaxation time mean value | Through study completion, an average of 6 months
Area under the ROC curve of the Apparent Diffusion Coefficient mean value | Through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Régional Universitaire de Nancy, Vandœuvre-lès-Nancy, France